CLINICAL TRIAL: NCT05794334
Title: Effects Of Low Dye Taping Technique Versus Robert Debre Method On Foot Posture And Range Of Motion In Children With Club Foot.
Brief Title: Low Dye Taping Technique Versus Robert Debre Method On Foot Posture And Range Of Motion In Children With Club Foot.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0738
Record Dates: First submitted 2023-02-20; First posted 2023-04-03 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Club Foot
Keywords: Low dye taping; Robert Debre tecnique
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dye Taping (Experimental): : There were 20 patients in group A which received the low dye taping technique. Low-dye is a classic taping method to reduces strain from plantar fascia and provide medial ankle arch support. If properly applied, reduces subtalar joint motion, pain, excessive pronation. Hence, it can be used in the treatment of ankle and foot.
  Interventions: Other: Low Dye Taping
- Robert Debre Method (Experimental): This second group also contains 20 participents.French functional method is similar to the Ponseti method. In this technique, the patient undergoes 30-minute daily session for 2 weeks and then twice a week until achieving foot correction. It consists of stretching of triceps surae to improve tibio-talar joint function. daily manipulations of the newborn's foot, stimulation and strenghtening of the muscles around the foot (particularly the peroneal muscles) and temporary immobilization of the foot with elastic and nonelastic adhesive taping so that the reduction achieved by.
  Interventions: Other: Low Dye Taping

INTERVENTIONS:
Other: Low Dye Taping — This second group also contains 20 participents.French functional method is similar to the Ponseti method. In this technique, the patient undergoes 30-minute daily session for 2 weeks and then twice a week until achieving foot correction. It consists of stretching of triceps surae to improve tibio-talar joint function. daily manipulations of the newborn's foot, stimulation and strenghtening of the muscles around the foot (particularly the peroneal muscles) and temporary immobilization of the foot with elastic and nonelastic adhesive taping so that the reduction achieved by.The average time of this method ranges between 6 to 8 weeks, with all the deformities being corrected apart from equinus. This method reports a 93% success rate
  Other Names: Robert Debre Technique

SUMMARY:
To Check the effects of the low dye taping technique versus the Robert Debre method on foot posture and range of motion in children with club feet.

DETAILED DESCRIPTION:
This study was a Randomized clinical trial. It was carried out in the physiotherapy department of children hospital Lahore,those patients were taken who had congenital clubfoot.40 patients were taken with the predetermined inclusive and exclusive criteria through non probability convenience sampling technique.All participants informed about the study,Group A received Low Dye taping Technique 2 times in a week for 6 weeks,while the group B received the Robert Debre Methpod daily 30 minutes session for total 6 weeks.Foot posture, range of motion and gait will be assessed by Demiglio bensahel and pirani scoring system with the help of goniometer and compared the results.Data analyzed by SPSS 25.0 statistical software. After checking the normality of data nonparametric tests applied to check the difference between and within the groups.

ELIGIBILITY:
Inclusion Criteria:

1. (1month to 6months ).
2. Children having idiopathic club foot
3. Unilateral or bilateral
4. Severity by Dimeglio Bensahel scale we include moderate ,severe and very severe feet

Exclusion Criteria:

1. Benign or non idiopathic.
2. An associated syndrome or neurological disease.
3. Positional club foot.
4. Those previously treated with another method in other hospitals.
5. Children with systemic diseases.
6. Juvenile Arthritis.

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-04-16 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
The Pirani scale: | 6th week
  The Pirani scale scoring system describes 6 signs of contracture with a three point scale: 0= no abnormality, 0.5= moderate abnormality, 1= severe abnormality. Scores for three midfoot signs (MFS) and three hindfoot signs (HFS), both with a maximum score of three are combined for a total score (TFS) out of six. Increasing scores indicates increasing severity, with zero indicating an unaffected foot and six the most severe clubfoot.
The Dimeglio Bensahel Classification: | 6th week
  The Dimeglio classification scores eight items; reducibility of four range of motion criteria and presence of four structural criteria. Reducibility of equinus, varus, midfoot rotation and midfoot adductus is scored zero to four points. The scores assigned to different degrees of reducibility of the deformity were specified by the author when the classification system was initially developed.The presence of four structural criteria; cavus, MC, PC, and muscle abnormality is also scored. Structural criteria are scored as 0= absent or 1= present. 8 Scores for the four reducibility criteria and the four structural criteria combine for an overall score, with 20 indicating the most severe clubfoot and zero an unaffected foot.

CONTACTS AND LOCATIONS:
Overall Officials: fareeha kausar, pp-Dpt, Principal Investigator — Riphah international university pakistan
Locations (1):
- Children hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No